CLINICAL TRIAL: NCT06560775
Title: Potential Effects of Nigella Sativa on T Lymphocytes and Inflammatory Cytokine Profile in Pediatric Systemic Lupus Erythematosus: A Randomized Controlled Trial
Brief Title: Effects of Nigella Sativa on T Cells and Cytokine Profile in Pediatric SLE Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brawijaya (Other)
Responsible Party: Principal Investigator, Wisnu Barlianto, Dr. dr. Wisnu Barlianto, Sp. A (K), Msi. med, University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SLE NS CBA
Record Dates: First submitted 2024-08-01; First posted 2024-08-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: SLE (Systemic Lupus)
Keywords: Immunomodulator; T lymphocyte; Inflammatory cytokine
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSO group (Experimental): NSO is 1 gram Nigella sativa oil in capsules. It was purchased from CV Rizki Abadi, Tuban East Java, Indonesia, with registration number POM TR. 183314171
  Interventions: Combination Product: Standard Treatment for SLE
- Placebo group (Placebo Comparator): Placebo capsules identical appearance contain 1 gram starch
  Interventions: Combination Product: Standard Treatment for SLE

INTERVENTIONS:
Combination Product: Standard Treatment for SLE — Standard Treatment for SLE

SUMMARY:
The goal of this clinical trial is to learn if Nigella sativa oil works to improve SLEDAI Score in SLE pediatric student. It will also learn about the Treg, T helper cells, and cytokine of the patient. The main questions it aims to answer are:

Does Nigella sativa oil lower the SLEDAI Score in pediatric patient? How does the effects of Nigella sativa oil on Treg cells, T helper cells, and cytokine in pediatric patient? Researchers will compare Nigella sativa oil group to a placebo group (a look-alike substance that contains no drug) to see if Nigella sativa oil works to treat SLE in pediatric patients.

Participants will:

Visit the clinic once in the beginning for pre treatment checkups. Take Nigella sativa oil or a placebo every day for 8 weeks. Visit the clinic once every 4 weeks for checkups. Visit the clinic after 8 weeks for post treatment checkups.

DETAILED DESCRIPTION:
SLE in paediatric patients requires long-term treatment with several side effects. Nigella sativa is known to have immunomodulatory effects. Our study aimed to investigate the immune-modulatory effects of Nigella sativa oil on T lymphocyte activity, inflammatory cytokine profile, and improvement of SLEDAI score in our patients. This was a placebo-controlled clinical trial of Nigella sativa oil administration in 32 paediatric SLE patients who were tested before and after treatment. The study subjects were randomly assigned. Patients had blood samples taken to be tested for T cell ratio, percentage of a number of cytokines (IFN-γ, TNF-α, IL-2, IL-4, IL-6, IL-17, and IL-10) using flow cytometry and CBA (Cytometric Bead Array), and SLEDAI score at the beginning of the study and after treatment. They were treated with 1 gram of N. sativa oil capsules and 1 gram of placebo daily for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric SLE patients aging between 1 and 18 years old according to the 2010 ACR-EULAR criteria
* Being under treatment with prednisone, hydroxychloroquine, and mycophenolic acid
* Not receiving any biological agent or cytokine inhibitors for at least 2 months prior to the intervention

Exclusion Criteria:

* Patients with any metabolic disorders (diabetes mellitus, Cushing's syndrome, and thyroid dysfunctions), any kidney or liver diseases, chronic inflammatory diseases (including inflammatory bowel diseases),
* Patients with history of taking antioxidant or anti-inflammatory supplements 2 months prior to the interventions

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
T cell lymphocyte and cytokine profiles, as well as SLEDAI Score | up to 4 months
  T cell lymphocyte includes Th1, Th2, Th17, and Treg in pg/mL (picograms per millilitre).
  Cytokine profiles includes IFN-γ, TNF-α, IL-2, IL-4, IL-6, IL-10, and IL-17α in pg/mL (picograms per millilitre).
  SLEDAI Score: SLE Disease Activity Index 2000 (SLEDAI-2K) in the point range between 0-105 (the higher the score the higher the disease activity). No activity (SLEDAI=0), mild activity (SLEDAI=1 to 5), moderate activity (SLEDAI=6 to 10), high activity (SLEDAI=11 to 19), and very high activity (SLEDAI≥20).
  T-cell lymphocytes and cytokine profiles will be used to determine the immunomodulating effect of Nigella sativa oil on the change of disease activity through the SLEDAI Score of paediatric SLE patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wisnu Barlianto, Dr. MD, Study Chair — Faculty of Medicine, Universitas Brawijaya; Desy Wulandari, MD, Study Director — Faculty of Medicine, Universitas Brawijaya; Tita L Sari, MD, Principal Investigator — Faculty of Medicine, Universitas Brawijaya; Rafika R Rachmaningrum, MD, Principal Investigator — Faculty of Medicine, Universitas Brawijaya; Rayi I Asasain, MD, Principal Investigator — Faculty of Medicine, Universitas Brawijaya
Locations (1):
- Universitas Brawijaya, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ciesielska-Figlon K, Wojciechowicz K, Wardowska A, Lisowska KA. The Immunomodulatory Effect of Nigella sativa. Antioxidants (Basel). 2023 Jun 24;12(7):1340. doi: 10.3390/antiox12071340. PMID 37507880
- [Result] Pop RM, Sabin O, Suciu S, Vesa SC, Socaci SA, Chedea VS, Bocsan IC, Buzoianu AD. Nigella Sativa's Anti-Inflammatory and Antioxidative Effects in Experimental Inflammation. Antioxidants (Basel). 2020 Sep 26;9(10):921. doi: 10.3390/antiox9100921. PMID 32993150
- [Result] Nasuti C, Fedeli D, Bordoni L, Piangerelli M, Servili M, Selvaggini R, Gabbianelli R. Anti-Inflammatory, Anti-Arthritic and Anti-Nociceptive Activities of Nigella sativa Oil in a Rat Model of Arthritis. Antioxidants (Basel). 2019 Aug 25;8(9):342. doi: 10.3390/antiox8090342. PMID 31450670
- [Result] Hikmah Z, Endaryanto A, Ugrasena IDG, Rahaju AS, Arifin S. Nigella sativa L. as immunomodulator and preventive effect on renal tissue damage of lupus mice induced by pristane. Heliyon. 2022 Apr 6;8(4):e09242. doi: 10.1016/j.heliyon.2022.e09242. eCollection 2022 Apr. PMID 35450390
- [Result] Kheirouri S, Hadi V, Alizadeh M. Immunomodulatory Effect of Nigella sativa Oil on T Lymphocytes in Patients with Rheumatoid Arthritis. Immunol Invest. 2016 May;45(4):271-83. doi: 10.3109/08820139.2016.1153649. Epub 2016 Apr 21. PMID 27100726
- [Result] Hadi V, Kheirouri S, Alizadeh M, Khabbazi A, Hosseini H. Effects of Nigella sativa oil extract on inflammatory cytokine response and oxidative stress status in patients with rheumatoid arthritis: a randomized, double-blind, placebo-controlled clinical trial. Avicenna J Phytomed. 2016 Jan-Feb;6(1):34-43. PMID 27247920

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT06560775/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT06560775/ICF_001.pdf